CLINICAL TRIAL: NCT03499782
Title: A Multi-center Study：Surgical Optimization and Prognosis Auxiliary System of Biliary Malignancies Based on Special Disease Database
Brief Title: Precise Treatment System of Biliary Malignancies Based on Special Disease Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shanghai Zhongshan Hospital (Other); Southwest Hospital, China (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Sun Yat-sen University (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Zhaohui Tang, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-JDYXY-2018-002
Record Dates: First submitted 2018-04-08; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Cholangiocarcinoma; Gall Bladder Carcinoma; Biliary System Disorder
Keywords: Prognosis; Surgery options; Bayesian networks
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Gallbladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malignant tumors of biliary system lack standard treatment and precise prognosis assessment methods. This study including 12 hospitals, collecting clinical and follow-up data of patients with biliary malignant tumors including cholangiocarcinoma and gallbladder carcinoma in recent 10 years, aim to build a special disease database, then use Bayesian networks and importance theory to establish a mathematical model to assess treatment strategies and prognosis accurately. At the same time, data on biliary malignant tumors newly treated by multicenters from 2018 to 2020 will be included to validate, adjust and refine the models to guide clinical individualized precise treatment.

ELIGIBILITY:
Inclusion Criteria：

* Clinical diagnosis of biliary malignancy including gallbladder carcinoma or cholangiocarcinoma verified by pathological results
* Must be able to undergo surgery
* Undergoing radical surgery for biliary malignancy (R0 or R1 resection)
* Not complicated with other malignancy
* No other treatments before and during surgery, such as radiotherapy and chemotherapy.

Exclusion Criteria:

* Non-primary gallbladder or cholangiocarcinoma
* With distant metastasis (M1 phase)
* Incomplete follow-up data
* Died within 30 days after surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Diagnosed with Gallbladder carcinoma or cholangiocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-05-25 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Death from biliary tract carcinoma | Every three months, up to five years
  Death from cholangiocarcinoma or gallbladder carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Geng, MD,PhD, Study Director — the first affiliated hospital of xi'an Jiaotong univerisity; Peng Gong, MD,PhD, Study Director — the first affiliated hospital of Dalian medical univerisity; Yu He, MD,PhD, Study Director — Southwest Hospital, China; Shengping Li, MD,PhD, Study Director — Cancer Institute and Hospital Affiliated to Sun Yat-sen University; Yinghe Qiu, MD,PhD, Study Director — Eastern Hepatobiliary Surgery Hospital; Zhi Dai, MD,PhD, Study Director — Shanghai Zhongshan Hospital; Tianqiang Song, MD,PhD, Study Director — Tianjin Medical University Cancer Institute and Hospital; Yudong Qiu, MD,PhD, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Jianying Lou, MD,PhD, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University; Jingdong Li, MD,PdD, Study Director — Affliated Hospital of North Sichuan Medical College; Wenlong Zhai, MD,PhD, Study Director — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Zhaohui Tang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided